CLINICAL TRIAL: NCT06921213
Title: Comprehensive Ambulatory Antibiotics for the Treatment of Congenital Syphilis
Acronym: Cares-1
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: University College Dublin (Other); University of Stellenbosch (Other); Malawi Liverpool Wellcome Programme (Other); University of Sydney (Other); Murdoch Childrens Research Institute (Other); MRC CTU at UCL (Unknown); PHPT/AMS Laboratory, Faculty of Associated Medical Sciences, Chiang Mai University (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 31732
Record Dates: First submitted 2025-03-25; First posted 2025-04-10 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-03

CONDITIONS: Syphilis, Congenital
MeSH Terms: conditions — Syphilis, Congenital | interventions — Linezolid; Amoxicillin; Penicillin G

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: It is not possible to blind the intervention to either participants or care providers given variation in route of administration and duration of therapy. Individuals assessing clinical and laboratory outcomes will be blinded to study group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Oral Linezolid (Experimental): 10 day course of Linezolid twice a day
  Interventions: Drug: Linezolid (LZD)
- Oral Amoxicillin (Experimental): 10 day course of Amoxicillin twice a day
  Interventions: Drug: Amoxicillin
- IM Benzathine penicillin (Active Comparator): Single IM dose of IM Benzathine penicillin
  Interventions: Drug: Benzathine Penicillin G

INTERVENTIONS:
Drug: Linezolid (LZD) — Ten day course. Oral Linezolid dosed at 10mg/kg twice a day.
  Arms: Oral Linezolid
Drug: Amoxicillin — Ten day course. Oral Linezolid dosed at 50mg/kg twice a day.
  Arms: Oral Amoxicillin
Drug: Benzathine Penicillin G — Single IM dose 50,000iu/kg
  Arms: IM Benzathine penicillin

SUMMARY:
CARES-1 is a randomised, open-label, phase II pharmacokinetic (PK) and safety study of ambulatory antibiotics for the treatment of neonates with "all-risk" asymptomatic congenital syphilis.

ELIGIBILITY:
Inclusion Criteria:

1. Infants at risk of congenital syphilis at birth defined as:

   1. an infant born to a mother who tests positive for syphilis in pregnancy using registered and licensed locally-available diagnostic tests for example but not limited to a Treponemal rapid POCT, an RPR or both.

      AND
   2. the mother is untreated in the current pregnancy defined as:

   i. she tested positive at antenatal care and received no treatment OR ii. she was never tested during antenatal care OR iii. she tested negative at antenatal care and positive on re-testing at delivery

   OR c. the mother is inadequately treated in the current pregnancy defined as:

   i. Having received a non-penicillin based treatment regimen; and/or ii. Does not have documentation of 3 doses of IM Benzathine Penicillin, given 7-10 days apart, with the last dose given > 30 days prior to delivery OR b. The mother was adequately treated in the current pregnancy BUT considers herself at risk of re-infection following a midwife delivered explanation of risk (partner treatment, multiple partners etc).
2. Infants who are asymptomatic for a diagnosis of congenital syphilis following application of a clinical proforma by the study team (Appendix 1)
3. Infants who are less than <= 7 days of life AND with a post-menstrual age (PMA) of 34-42 weeks (Appendix 2).
4. Infants who are tolerating enteral feeds, including if they are being administered by an NG tube.

Exclusion Criteria:

- 1. The infant's clinical condition at birth or prior to randomisation requires ongoing (> 48 hours) treatment with antibiotics with the potential for anti-treponemal activity i.e. B-lactams, Cephalosporins, Carbapenems.

2. They have a birthweight <2kg 3. They are nil by mouth. 4. They have a life-limiting congenital anomaly

Ages: 0 Days to 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Time above MIC in serum | From enrolment through to day 10 of the study
  Time above MIC of T. pallidum for the dosing interval in serum
Time above MIC in CSF | 10 days
  Time above MIC in CSF throughout the dosing interval
Adverse Events | Assessed from enrolment through to 24 weeks
  The proportion of individuals experiencing an adverse event through to week 24. The trial will record SAE, SUSARS, and drug related AEs of grade 3 or higher.

SECONDARY OUTCOMES:
Clinical Outcome | Enrolment through to week 24
  Proportion of infants who have clinical or laboratory evidence of congenital syphilis as adjudicated by an expert committee, blinded to treatment allocation, based on clinical and laboratory data.
AUC/MIC Ratio in serum | Enrolment through to day 10
  Proportion of individuals achieving an AUC/MIC ratio ≥100 in serum
AUC/MIC Ratio in CSF | Enrolment through to day 10
  Proportion of individuals achieving an AUC/MIC ratio ≥100 in CSF

CONTACTS AND LOCATIONS:
Overall Officials: Michael Marks, Principal Investigator — London School of Hygiene and Tropical Medicine; Bridget Freyne, Principal Investigator — University College Dublin
Locations (3):
- Universitas Indonesia, Jakarta, Indonesia
- Malawi Liverpool Wellcome Programme, Blantyre, Malawi
- Stellenbosch, Stellenbosch, South Africa

IPD SHARING:
Plan to Share IPD: Yes
At completion of the study an anonymised dataset will be deposited in an appropriate repository to facilitate sharing of IPD.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Following completion of the study
Access Criteria: Data will be available via a repository to other researchers